CLINICAL TRIAL: NCT00375037
Title: Cluster Randomized Controlled Trial of a Multifaceted Intervention to Improve Hand Hygiene Among Healthcare Workers
Brief Title: A Multifaceted Intervention to Improve Hand Hygiene
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05-277
Record Dates: First submitted 2006-09-11; First posted 2006-09-12 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Handwashing; Infection
Keywords: hand washing; cluster randomized trial; performance feedback; healthcare workers; Hand hygiene; hand washing adherence
MeSH Terms: conditions — Infections | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hand hygiene (Experimental): Hand hygiene promotion
  Interventions: Behavioral: feedback; Behavioral: Education
- Usual care (Active Comparator): usual care
  Interventions: Other: usual care

INTERVENTIONS:
Behavioral: feedback
  Arms: Hand hygiene
Behavioral: Education
  Arms: Hand hygiene
Other: usual care
  Arms: Usual care

SUMMARY:
This randomized controlled trial will evaluate the effect of a multifaceted intervention including performance feedback on adherence to hand hygiene among healthcare workers. A key component of the study is to demonstrate whether improved adherence to hand hygiene leads to a reduction in rates of infection.

DETAILED DESCRIPTION:
A cluster randomized controlled trial of the intervention will be conducted where hospital units (wards) in three hospitals will be allocated to either the intervention or usual practise. We will stratify by hospital site in order to minimize confounding by hospital-level factors. The unit of allocation, intervention, and analysis will be at the level of the hospital unit. Thirty hospital units will be randomized to either the intervention or comparison arm. We will compare adherence to hand hygiene, MRSA rates, and other outcomes between the two study arms.

ELIGIBILITY:
A. Study units Inclusion: Medical and subspecialty units, surgical units, critical care units

Exclusion: pediatric units, neonatal intensive care units

B. Healthcare workers

Inclusion: any hospital staff with direct patient care who are affiliated with a single unit (includes registered nurses, nursing assistants, environmental aides, allied health professionals (occupational, physical, and respiratory therapists), and some physicians

C. Patients Clinical outcomes will be measured in patients on study units.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2007-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Incidence of MRSA | 12 months
Adherence to hand hygiene | 12 months

SECONDARY OUTCOMES:
Incidence of multi-resistant bacteria other than MRSA | 12 months
Catheter-related blood stream infections | 12 months
Clostridium difficile related diarrhea | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Loeb, MD, MSc, Principal Investigator — Hamilton Health Sciences- McMaster University
Locations (3):
- Canada (3):
  - Hamilton General Hospital, Hamilton, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - Henderson Hospital, Hamilton, Ontario